CLINICAL TRIAL: NCT04344899
Title: Pediatric Oncology Recovery Trial After Surgery
Acronym: PORTS
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0964.cc; NCI-2021-10775 (Other: CTRP)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Cancer
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Historical: Retrospective Review
  Interventions: Other: Observational
- ERAS Patients: Prospective Review
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Enhanced Recovery After Surgery protocol at five tertiary-care pediatric hospitals in pediatric patients undergoing abdominal or retroperitoneal surgical resections for cancer.
  Other Names: ERAS Protocol

SUMMARY:
Pediatric Oncologic Recovery Trial After Surgery (PORTS) trial is an investigator-initiated, multicenter, multidisciplinary prospective case-control study of the implementation of an Enhanced Recovery After Surgery (ERAS) protocol at five tertiary-care pediatric hospitals in pediatric patients undergoing abdominal or retroperitoneal surgical resections for cancer. A pilot phase will determine characteristics of a successful protocol implementation and an exploratory phase plans to examine adherence, objective patient outcomes, and patient-reported outcomes. After completing primary enrollment, this collaborative will continue to enroll patients in the shared data registry and continue to refine the underlying ERAS protocol developed for this project.

DETAILED DESCRIPTION:
Two arms:

Historical patients ERAS patients

Number of patients: 288

Primary outcome

· Number of 90-day complications by Clavien-Dindo classification

Secondary outcome(s):

* Adherence to ERAS protocol items with # of items achieved (out of 20)
* Length of stay
* Re-admissions within 90 days
* Re-operations within 90 days
* Number of visits to the emergency room within 90 day period
* Minimum, mean, maximum daily pain score during first 7 days after surgery
* Mean daily IV morphine equivalents (mg/kg) usage during first 7 days after surgery

  * recurrence free survival (months)
  * overall survival (months)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing operations at a pediatric hospital setting aged 1 month or older
* Parents of patients undergoing operations at pediatric hospital settings aged 1 month or older
* Undergoing urologic reconstruction, ureteral operations, pyeloplasty, intraabdominal on-cologic resections, urachal remnant excision, bariatric operations, pectus surgery, ap-pendicitis, orthopedic or neurosurgical operations and inflammatory bowel disease proce-dures
* Providers of patients undergoing surgery in pediatric settings

Exclusion Criteria:

* Less than 1 month in age

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing urological surgery
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of 90-day complications by Clavien-Dindo classification | 90 Days

SECONDARY OUTCOMES:
Number of Adherence issues to ERAS protocol items with # of items achieved (out of 20) | 90 Days
Length of stay | 90 Days
Number of Re-admissions within 90 days | 90 Days
Number of Re-operations within 90 days | 90 Days
Number of visits to the emergency room within 90 day period | 90 Days
VAS daily pain score during first 7 days after surgery | 90 Days
Mean daily IV morphine equivalents (mg/kg) usage during first 7 days after surgery | 90 Days
Recurrence free survival (months) | 90 Days
Overall survival (months) | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Rove, MD, Principal Investigator — Childrens Hospital Colorado
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansfield SA, Kotagal M, Hartman S, Murphy AJ, Davidoff AM, Anghelescu DL, Mecoli M, Cost N, Hogan B, Rove KO. Development of an enhanced recovery after surgery program for pediatric solid tumors. Front Surg. 2024 May 22;11:1393857. doi: 10.3389/fsurg.2024.1393857. eCollection 2024. PMID 38840973